CLINICAL TRIAL: NCT05853354
Title: A Randomized, Double-blind, Parallel-group, Active-controlled Comparative Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Immunogenicity of LY06006 Compared With EU-Prolia in Postmenopausal Women With Osteoporosis
Brief Title: Comparative Efficacy, Safety, PK, and Immunogenicity Study
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: LY06006/MRCT-301; IND 138591 (Registry Identifier: FDA); 2022-002312-23 (EudraCT Number)
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Comparative efficacy;safety;PK; immunogenicity; biosimilar
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, parallel-group, active-controlled, comparative study (Main Period) with a Transition Period to compare the efficacy, PD, safety, PK and immunogenicity of LY06006 and EU-Prolia among female participants with postmenopausal osteoporosis.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Upon enrollment, each participant will receive a unique participant identification number.Participant numbers must not be re-used for any other participants.
  Prior to dosing in the Transition Period and to maintain the blind throughout the study, participants will be re-randomized and receive a second randomization number. Participants randomized to receive EU-Prolia in the Main Period will be re-randomized to receive either LY06006 or continue to receive EU-Prolia. Participants who received LY06006 in the Main Period will be re-randomized to continue to receive LY06006 in the Transition Period. All participant assignment during the Transition Period will be performed via the IRT system to maintain the blind of treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY06006 (Experimental): to be administered 2 doses to the patients at the main treatment period and 1 dose at the transition period.
  Interventions: Biological: Denosumab
- EU Prolia (Active Comparator): to be administered 2 doses to the patients at the main treatment period and 1 dose at the transition period.
  Interventions: Biological: Denosumab

INTERVENTIONS:
Biological: Denosumab — Sterile, preservative-free, solution of denosumab packed in 1-mL pre-filled glass syringes for subcutaneous administration.Each syringe contains 60 mg denosumab (60 mg/mL solution) and is intended for single administration once every 6 months.

SUMMARY:
this comparative clinical study is designed to demonstrate that LY06006 and EU-Prolia have no clinically meaningful differences in clinical efficacy, pharmacodynamic (PD), safety, PK, and immunogenicity in postmenopausal women with osteoporosis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel-group, active-controlled, comparative study (Main Period) with a Transition Period to compare the efficacy, PD, safety, PK, and immunogenicity of LY06006 and EU-Prolia among female participants with postmenopausal osteoporosis.

Participants will go through a Screening Period within 35 days prior to first dosing. After signing the informed consent form (ICF), participants will be screened for age, menopausal status, and vitamin D levels, in addition to other inclusion/exclusion criteria. Participants will also undergo a screening DXA examination. Eligibility is based on the absolute value consistent with a T-score ≤ -2.5 and ≥ -4.0 at the lumbar spine.

Main Period Upon completing all screening assessments and meeting all eligibility criteria, participants will enter the Main Period of the study. The Main Period will last 12 months where participants will be randomized in a 1:1 ratio to receive either a dose (60 mg/1 mL) of LY06006 or EU-Prolia subcutaneously at the Baseline Visit (Day 1) and Month 6. All participants will receive daily supplements of elemental calcium (at least 1000 mg) and vitamin D (at least 400 IU). Study visits will occur at the Baseline Visit (Day 1), and at Months 0.5, 1, 2, 3, 6, 9, and 12.

Follow-up BMD assessment will be done at Months 6 and 12. Blood sampling for PD, safety, PK, and immunogenicity will be done at the Baseline Visit (Day 1), and at Months 0.5, 1, 2, 3, 6, 9, and 12.

Transition Period The Transition Period will be conducted in all participants who completed the Main Period of the study. At Month 12, participants who received EU-Prolia in the Main Period will be re-randomized in a 1:1 ratio to either be transitioned to receive a dose of LY06006 or continue on EU-Prolia subcutaneously. Participants who received LY06006 in the Main Period will be re-randomized to continue to receive LY06006 in the Transition Period. All participant assignment during the Transition Period will be performed via the interactive response technology (IRT) system to maintain the blind of treatment assignment.

Blood sampling for PD, safety, PK, and immunogenicity will be done at Months 15 (PK and immunogenicity only) and 18. End of study (EoS) assessments will be performed at Month 18 or at the time of early discontinuation or withdrawal of the participant. The duration of the clinical phase for participants from the Screening Period until the EoS Visit is approximately 19 months (up to 5 weeks of Screening Period, 12 months of Main Period, and 6 months of Transition Period).

ELIGIBILITY:
Inclusion Criteria:

Age

1. Participant is ≥ 60 to ≤ 90 years of age inclusive, at the time of signing the informed consent.

   Type of Participant and Disease Characteristics
2. Participant is an ambulatory postmenopausal woman (defined as lack of menstrual period for at least 12 months prior to Screening Visit, for which there is no other obvious pathological or physiological cause).

   * Serum FSH test can be done at the Screening Visit in case of uncertainty.
   * Female participants who underwent bilateral oophorectomy (with or without hysterectomy) at least 6 weeks prior to the Screening Period are eligible to participate.
3. Participant is diagnosed with osteoporosis, with absolute BMD consistent with a T-score of ≤ -2.5 and ≥ -4.0 at the lumbar spine (L1-L4 region) as measured by DXA at the Screening Visit.
4. Participant has at least two lumbar vertebrae in L1-L4 region and one hip evaluable by DXA for BMD measurement at the Screening Visit.

Weight 5. Participant has body weight ≥ 50 kg and ≤ 90 kg at Screening. Informed Consent 6. Participant is able to read and understand, and willing to provide signed informed consent as described in Appendix 1, Section 10.1.3 which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

-

Exclusion Criteria:

Medical Conditions

1. Participant has a history and/or presence of any severe or more than two moderate vertebral fractures as determined by central reading of lateral spine X-ray at Screening Visit.
2. Participant has a history and/or presence of hip fracture.
3. Participant has a history and/or presence of atypical femur fracture.
4. Participant presents with any active healing fracture, per assessment of the Investigator.
5. Participant has a history of bilateral hip replacement (unilateral is allowed if the other hip is evaluable by DXA).
6. Participant has history and/or presence of osteonecrosis of the external auditory canal.
7. Evidence of any of the following conditions which may affect BMD or interfere with the interpretation of the findings:

   1. Participant has a history of bone disease e.g., osteomalacia, osteopetrosis, Paget's disease, or osteogenesis imperfecta.
   2. Participant has a history of metabolic or other endocrinologic diseases such as Cushing's disease, hyperprolactinemia, hypopituitarism, acromegaly, malabsorption syndrome (or any gastrointestinal disorders associated with malabsorption, e.g., Crohn's disease and chronic pancreatitis).
   3. Participant has a history of chronic inflammatory diseases, obvious sclerosis, osteophytosis, severe scoliosis, or other degenerative changes due to other co-morbidities.
   4. Participant has a history or current hyperparathyroidism or hypoparathyroidism. Note: Mild non-clinically significant secondary hyperparathyroidism may be acceptable upon discussion with the Medical Monitor.
   5. Participant has current uncontrolled hyperthyroidism or hypothyroidism. Note: Participants with hypothyroidism who are on stable thyroid hormone replacement therapy may be allowed per the following criteria:

      * If TSH level is within normal range, the participant is eligible.
      * If TSH level is elevated (> 5.5 μIU/mL and ≤ 10.0 μIU/mL) and serum free T4 is within normal range, the participant is eligible. If TSH is below the lower level of normal, the participant should be excluded.
   6. Participant has other disease conditions where there is bone/joint involvement (e.g., rheumatoid arthritis, ankylosing spondylitis, gout, multiple myeloma, achondroplasia, bone metastases, renal osteodystrophy, osteomyelitis).
8. Participant has hypocalcemia (defined as albumin adjusted serum calcium level < 2.0 mmol/L [8.0 mg/dL] Grade 2 per Common Terminology Criteria for Adverse Events version 5.0) or hypercalcemia (defined as albumin adjusted serum calcium levels > 2.62 mmol/L [10.50 mg/dL]).
9. Participant has vitamin D deficiency (defined as 25-hydroxy vitamin D level < 20 ng/mL [< 50 nmol/L]).

   Note: Oral replenishment of vitamin D is permitted at the discretion of the Investigator and in accordance with local standard of care during the Screening Period. Participants can be enrolled if a repeat test (post supplementation) prior to enrollment shows corrected 25-hydroxy vitamin D level ≥ 20 ng/mL (≥ 50 nmol/L).
10. Participant has any malignancy (except fully resected cutaneous basal cell or squamous cell carcinoma, cervical or breast ductal carcinoma in situ) within the last 5 years.
11. Participant has known history of liver cirrhosis.
12. Participant has known history of hepatitis B, hepatitis C, or HIV infection, or an active infection including, but not limited to SARS-CoV-2, tests positive for hepatitis B (positive HBsAg, positive anti-HBc with negative anti-HBs), hepatitis C (hepatitis C antibody), or HIV antibody during the Screening Period.
13. Participant has oral or dental conditions:

    1. Prior history or current evidence of osteomyelitis or osteonecrosis of the jaw.
    2. Active dental or jaw condition which requires oral surgery.
    3. Invasive dental procedure planned during the study or within the past 6 months (e.g., tooth extraction, dental implants, oral surgery).
    4. Non-healed dental or oral surgery.
    5. Active periodontal disease.
    6. Poor oral hygiene.
14. Participant has a history of major surgery within 8 weeks prior to the Screening Period or planned, anticipated major surgery during the study.
15. Participant has a history and/or presence of significant cardiac disease or ECG abnormalities indicating significant risk for participating in the study as judged by the Investigator.

    Prior/Concomitant Therapy
16. Participant shows contraindications to denosumab therapy (e.g., hypocalcemia), or calcium or vitamin D supplementation before starting study intervention administration.
17. Participant requires ongoing use of any osteoporosis treatment (other than calcium and vitamin D supplements).
18. Use of any of the below medications that can affect BMD:

    l. Denosumab used at any time prior to Screening Visit.
    1. Oral bisphosphonates at any dose for osteoporosis treatment:

       * Used for > 3 years cumulatively at Screening Visit.
       * At any dose used within 1 year prior to Screening Visit (if ≤ 3 years of use cumulatively).
    2. Intravenous bisphosphonate at any dose within 5 years prior to Screening Visit.
    3. PTH or PTH analogues at any dose within 2 years prior to Screening Visit.
    4. Systemic HRT (oral or transdermal estrogen), SERMs, tibolone, aromatase inhibitors, or androgens at any dose within 1 year prior to Screening Visit.

       Note: Exceptionally, non-systemic vaginal estrogen treatment is permitted.
    5. Calcitonin, or its derivatives, and calcimimetics (such as cinacalcet or etelcalcetide) at any dose within 12 months prior to Screening Visit.
    6. Calcitriol, alfacalcidol, or eldecalcitol within 3 months of the Screening Visit.
    7. Fluoride or strontium at any dose at any time prior to Screening Visit.
    8. Romosozumab or cathepsin K inhibitors received at any time prior to Screening Visit.
    9. Systemic glucocorticoids (≥ 5 mg prednisone or equivalent per day for more than 10 days or cumulative ≥ 50 mg) within 3 months prior to Screening Visit.
    10. Other bone active drugs including anticonvulsants (except benzodiazepines, gabapentin, and pregabalin), heparin (including low molecular weight heparins), vitamin K (supplementation or therapeutic dose), vitamin K antagonists (e.g., warfarin, acenocumarol), emtricitabine, tenofovir, adefovir, systemic ketoconazole, adrenocorticotropic hormone, lithium, protease inhibitors, gonadotropin-releasing hormone agonist, aluminum, barbiturate, methotrexate, chemotherapeutic agents, cyclosporine, tacrolimus, or anabolic steroids at any dose within 3 months prior to Screening Visit. Prior/Concurrent Clinical Study Experience
19. Participant is receiving or has received another investigational product within 1 month or 5 half-lives of the other investigational product, whichever is longer, before study intervention administration in this study. Diagnostic Assessments
20. Participant has DXA measurements where:

    1. Height, weight, or girth measurements may preclude accurate DXA measurements in the Investigator's opinion.
    2. BMD absolute value is consistent with a T-score < -4.0 at the total hip or femoral neck.
21. Participant has severe renal impairment (defined as participant in dialysis or with an eGFR < 30 mL/min per MDRD formula).
22. Participant has inadequate hepatic function (ALT and/or AST ≥ 2 × ULN).
23. Participant presents with clinically significant leukopenia, neutropenia, or anemia as judged by the Investigator.

    Other Exclusion Criteria
24. Participant has a known intolerance to calcium or vitamin D supplements.
25. Participant has a history of prescription drug abuse or any illicit drug use within 6 months prior to Screening Visit.
26. Participant has a history of alcohol abuse (defined as consuming more than 3 drinks on any day or more than 7 drinks per week) according to medical history within 6 months prior to Screening Visit.
27. Participant is a smoker or has used nicotine and nicotine-containing products within 12 months of Screening Visit.
28. Participant has a known sensitivity to mammalian cell-derived drug products.
29. Participant is immunosuppressed for any reason.
30. Participant has any other conditions including clinically significant medical conditions/disorders/diseases, psychiatric status, or laboratory abnormalities that in the opinion of the Investigator might interfere with the participant's ability to participate in the study, would pose a risk to the participant's safety, or interfere with the study evaluation, procedure, or completion.

Ages: 60 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — lack of menstrual period for at least 12 months prior to Screening Visit, for which there is no other obvious pathological or physiological cause
Enrollment: 392 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To demonstrate equivalent efficacy between LY06006 and EU-Prolia, in terms of BMD in female participants with postmenopausal osteoporosis; | 12 months
  %CfB in lumbar spine BMD at Month 12
EU Marketing Authorization only: To demonstrate similar PD between LY06006 and EU-Prolia, in terms of the bone resorption marker sCTX in female participants with postmenopausal osteoporosis | 6 months
  EU Marketing Authorization only: standardized AUEC0-6m (post first dose) of -%CfB in bone resorption marker sCTX over 6 months

SECONDARY OUTCOMES:
To provide additional comparative efficacy data of LY06006 with EU-Prolia in female participants with postmenopausal osteoporosis | 6-12 months
  * %CfB in lumbar spine BMD at Month 6
  * %CfB in total hip BMD at Months 6 and 12
  * %CfB in femoral neck BMD at Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Joe Tai, Study Chair — Luye Pharma Group Ltd.
Locations (38):
- United States (3):
  - Clinical Trials Management Services, LLC, Thousand Oaks, California
  - Indago Research and Health Center, Inc., Hialeah, Florida
  - Valley Institute of Research, Fort Worth, Texas
- Bulgaria (4):
  - MHAT Dr. Atanas Dafovski AD, Kardzhali
  - Medical Centre Leo Clinic EOOD, Plovdiv
  - Diagnostic-consultative center Ascendent EOOD, Sofia
  - Medical Center Leo Clinic EOOD, Varna
- Czechia (2):
  - CCR Brno s.r.o., Brno
  - Synexus Prague, Prague
- Japan (11):
  - Gifu Prefectural General Med C., Gifu, Gihu
  - Asakawa Orthopedic Clinic, Chikugo, Hukuoka
  - Obase Hospital - Orthopedics, Miyako-gun, Hukuoka
  - Himeno Hospital, Yame-gun, Hukuoka
  - Marunouchi Hospital, Matsumoto-shi, Nagano
  - Nemoto Geka SeikeiGeka, Fujimi, Saitama
  - Kobayakawa Orthopedic Rheumatologic, Fukuroi, Shizuoka
  - Med Teda Ooimachi Orthopaedic, Shinagawa-ku, Tôkyô
  - Koenji Orthopedic Surgery, Shinagawa-ku, Tôkyô
  - Shimonoseki City Hospital, Shimonoseki, Yamaguchi
  - Nakamura Hospital, Beppu, Ôita
- Poland (18):
  - Centrum Medyczne Pratia Poznan, Skórzewo, Greater Poland Voivodeship
  - Synexus Polska Sp. z o.o., Katowice, Silesian Voivodeship
  - Centrum Medyczne Pratia Czestochowa, Częstochowa
  - Synexus Polska Sp. z o.o., Częstochowa
  - Synexus Polska Sp. z o.o., Gdansk
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Pratia Jelenia Gora, Jelenia Góra
  - Centrum Medyczne Pratia Katowice, Katowice
  - Pratia MCM Krakow, Krakow
  - Krakowskie Centrum Medyczne Sp.z o.o., Krakow
  - Synexus Polska Sp. z. o.o., Lodz
  - Centrum Medyczne AMED Oddzial w Lodzi, Lodz
  - Synexus Polska Sp. z o.o., Poznan
  - FutureMeds Warszawa Centrum, Warsaw
  - Synexus Polska Sp. z o.o., Warsaw
  - Centrum Medyczne AMED, Warsaw
  - Synexus Polska Sp. z o.o., Wroclaw
  - FutureMeds Sp. z o.o., Wroclaw